CLINICAL TRIAL: NCT02688894
Title: The Molecular Screening Study for the Umbrella Trial (SUKSES) in Relapsed Small Cell Lung Cancer Patients [SUKSES-S]
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Se-Hoon Lee, MD,PhD, Samsung Medical Center
Other Study IDs: 2016-02-071
Record Dates: First submitted 2016-02-18; First posted 2016-02-23 (Estimated); Last update posted 2024-01-03 (Actual); Status verified 2023-12

CONDITIONS: Small Cell Lung Cancers; Neuroendocrine Carcinoma
MeSH Terms: conditions — Carcinoma, Neuroendocrine

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Tumor tissue, whole blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Small cell lung cancers: To provide molecular characteristics of Small cell lung cancers to proceed SUKSES trial, To assess success rate of molecular profiling of Small cell lung cancers
  Interventions: Other: No treatment is included in this protocol.

INTERVENTIONS:
Other: No treatment is included in this protocol. — Tumor tissues (fresh or archival) will be analyzed using NGS-based cancer panel, nanostring CNV, immunohistochemistry and/or FISH.
  Specific methods of each molecular tests will be defined with standard laboratory manual developed by pathologists.

SUMMARY:
This protocol is a molecular screening protocol only. No drug intervention study will be included in this protocol. Based on the molecular profiling, patients may be eligible for drug intervention study of SUKSES trial.

This procedure can be performed during or after the first-line treatment. DNA will be extracted from the archived or fresh tissue and blood. NGS-based cancer panel and Nanostring CNV will be tested with DNA from tissue and/or blood.

Immunohistochemistry and FISH will be done by pathologists using archived or fresh tissue.

Tumor tissues (fresh or archival) will be analyzed using NGS-based cancer panel, nanostring CNV, immunohistochemistry and/or FISH.

Specific methods of each molecular tests will be defined with standard laboratory manual developed by pathologists.

DETAILED DESCRIPTION:
This protocol is a molecular screening protocol only. No drug intervention study will be included in this protocol. Based on the molecular profiling, patients may be eligible for drug intervention study of SUKSES trial.

This procedure (molecular profiling) can be performed before, during, or after the initial treatment.

DNA will be extracted from the archived or fresh tissue and blood. NGS-based cancer panel and Nanostring CNV will be tested with DNA from tissue and/or blood.

Immunohistochemistry and FISH will be done by pathologists using archived or fresh tissue.

In addition, blood collection will be conducted at Baseline (initial), three weeks, six weeks, twelve weeks, and subsequent imaging.

Tumor tissues (fresh or archival) will be analyzed using NGS-based cancer panel, nanostring CNV, immunohistochemistry and/or FISH. Specific methods of each molecular tests will be defined with standard laboratory manual developed by pathologists.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of fully informed consent prior to any study specific procedures.
2. Patients must be ≥20 years of age.
3. Histologically or cytologically confirmed Small cell lung cancers
4. ECOG performance status of 0 to 2
5. Patients who are being treated or were treated with platinum-based chemotherapy as a first-line treatment
6. Patients with available archival tissues for molecular analysis or patients who agreed with biopsy for molecular analysis

Exclusion Criteria:

1. More than two prior chemotherapy regimen for the treatment of small cell lung cancer
2. Pregnant or nursing women (women of reproductive potential have to agree to use an effective contraceptive method)
3. Patients with second primary cancer, except: adequately treated non-melanoma skin cancer, curatively treated in-situ cancer of the cervix, or other solid tumours curatively treated with no evidence of disease for ≤2 years.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Histologically or cytologically confirmed Small cell lung cancers
Sampling Method: Probability Sample
Enrollment: 797 (Estimated)
Dates: Start 2016-04-29 (Actual); Primary Completion 2024-09 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Ratio of each molecular subtypes | After registration of this study
  To provide molecular characteristics of SCLC to proceed SUKSES trial

SECONDARY OUTCOMES:
Success rate of each molecular profiling methods | After completion of registration
  To provide molecular characteristics of SCLC to proceed SUKSES trial

CONTACTS AND LOCATIONS:
Overall Officials: Se-Hoon Lee, MD, PhD, Principal Investigator — Samsung Medical Center
Locations (6):
- South Korea (6):
  - Gachon University Gil Medical Center, Incheon
  - Chungbuk University Hospital, Jungbuk
  - Seoul National University Bundang Hospital, Seongnam
  - Samsung Medical Center, Seoul
  - VHS Medical Center, Seoul
  - Ulsan University Hospital, Ulsan